CLINICAL TRIAL: NCT02036684
Title: A Multicentre, Pilot Randomized Controlled Trial to Examine the Effects of Prehabilitation on Functional Outcomes After Radical Prostatectomy
Brief Title: Prehabilitation for Prostate Cancer Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Guelph-Humber (Other)
Collaborators: University Health Network, Toronto (Other); Princess Margaret Hospital, Canada (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Daniel Santa Mina, Program Head, University of Guelph-Humber
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: D-201327
Record Dates: First submitted 2013-11-16; First posted 2014-01-15 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer Patients Undergoing Radical Prostatectomy
Keywords: Prostate cancer; Radical prostatectomy; Prehabilitation; Pelvic floor muscle exercises
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Lifestyle Booklet (No Intervention): Standard care for radical prostatectomy (RP) patients includes the provision of preoperative information from a urology nurse educator. Usual care (UC) participants will be given generic instructions by the research coordinator about pelvic floor muscle exercises (PFMX), mobilization and general timeframes for a return to normal activities. The UC group will receive the same PFMX prescription as the PREHAB (Experimental) group and will receive weekly communication from the research coordinator regarding compliance with the PFMX prescription to provide an attentional-control. These instructions are provided in a healthy lifestyle booklet for men with prostate cancer.
- Prehabilitation (PREHAB) (Experimental): The prehabilitation (PREHAB) program focuses on total-body physical exercises and pelvic floor muscle exercises (PFMX). The total-body exercise prescription will consist of 60 minutes of home-based, unsupervised exercise on 3-4 days per week, alternating between aerobic and resistance training. Each session will include: a 5-minute warm-up, 25 minutes of aerobic exercise, 25 minutes of resistance training (5 exercises targeting major muscle groups), and a 5-minute cool-down. Training intensity progression will occur throughout the intervention. Participants will be provided with resistance bands, a stability ball, and an exercise mat. The PFMX prescription will include a gradual increase in PFMX exercises from 60 per day during weeks 1-2, 120 per day during weeks 3-4, and 180 per day during weeks 5-6 until the surgery date. The total number of repetitions of the PFMXs will be divided equally between the rhythmic and sustained contractions.
  Interventions: Behavioral: Prehabilitation (PREHAB)

INTERVENTIONS:
Behavioral: Prehabilitation (PREHAB)
  Arms: Prehabilitation (PREHAB)

SUMMARY:
Radical prostatectomy is the most common and effective treatment for localized prostate cancer. Unfortunately, radical prostatectomy is associated with significant adverse effects, such as urinary incontinence, sexual dysfunction, and reduced physical function that collectively diminish health-related quality of life which may persist for up to two years postoperatively. The primary objective of this trial is to assess the feasibility of conducting of a multi-site randomized controlled trial to test the effect of a comprehensive prehabilitation program versus standard care for men with prostate cancer undergoing radical prostatectomy. We hypothesize that men with prostate cancer undergoing radical prostatectomy in the comprehensive prehabilitation program (full-body exercises and pelvic floor muscle exercises) will report better health-related quality of life, urological symptoms, and physical fitness, physical activity, and pain, as well as a shorter postoperative length of stay than participants receiving standard preoperative care (pelvic floor muscle exercises alone). Our secondary objective is to report estimates of efficacy on several clinically important outcomes for this population that will be used for sample size calculations in an adequately powered trial.

ELIGIBILITY:
Inclusion Criteria:

* Men with localized prostate cancer (stage cT1- cT2) who have consented for radical prostatectomy
* between the ages of 40 and 80 years.

Exclusion Criteria:

* i) severe coronary artery disease (Canadian Cardiovascular Society class III or greater);
* ii) significant congestive heart failure (New York Heart Association class III or greater);
* iii) uncontrolled pain;
* iv) neurological or musculoskeletal co-morbidity inhibiting exercise;
* v) diagnosed psychotic, addictive, or major cognitive disorders;
* vi) no more than two of the following Coronary Risk Factors as defined by the American College of Sports Medicine : family history of coronary disease, cigarette smoking, hypertension (SBP > 140 mmHg; DBP > 90 mmHg), known dyslipidemia, known impaired fasting, glucose (>110 mg/dL), obesity (BMI > 30 kg/m2 or waist circumference > 102cm), or physically inactive (<150 min of moderate intensity physical activity per week).

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05-17 (Actual); Study Completion 2016-05-17 (Actual)

PRIMARY OUTCOMES:
Recruitment | When recruitment is complete (approximately 12 months after study initiation; January 2015)
  Prior exercise trials in prostate cancer patients on hormone and/or radiation therapy have observed recruitment rates of 25-40%, but no studies have assessed recruitment to a preoperative exercise intervention among prostate cancer survivors. We will measure recruitment-success percentage and will record reasons for non-participation to better understand why men electing radical prostatectomy would not participate in an exercise intervention.
Adherence to Prehabilitation Program | 26 weeks postoperatively
  Adherence to the home-based exercise program (aerobic and resistance) and pelvic floor muscle exercises will be measured through a logbook completed by the research coordinator during weekly communication.
Contamination | 26 weeks postoperatively
  The same exercise logbook questions that ask about aerobic and resistance exercise, and pelvic floor muscle exercises, will be administered to both groups to assess contamination.
Study Retention | 26 weeks postoperatively
  Retention will be assessed by measuring attrition throughout the intervention period and at each assessment.

SECONDARY OUTCOMES:
Physical Fitness | At baseline, within 1 week prior to surgery, and at 4, 12, and 26 weeks postoperatively.
  Musculoskeletal fitness will be assessed using grip strength (hand dynamometer) and maximal upper body strength (handheld digital dynamometer). Body composition will be assessed via body mass index, waist circumference (midpoint between lowest rib and iliac crest), and body fat percentage (bioelectrical impedance analysis). Aerobic fitness is measured using the 6-Minute Walk Test.
Quality of Life | At baseline, within 1 week prior to surgery, and at 4, 12, and 26 weeks postoperatively.
  Prostate cancer-specific health related quality of life (HRQOL) will be measured using the Functional Assessment of Cancer Treatment-Prostate (FACT-P) and the Patient-Oriented Prostate Utility Scale (PORPUS).
Psychosocial Wellbeing | At baseline, within 1 week prior to surgery, and at 4, 12, and 26 weeks postoperatively.
  Depressive symptoms will be measured with the 14-item Hospital Anxiety and Depression Scale (HADS). Cancer-specific fatigue will be measured using the FACT-Fatigue which is a widely used 13-item measure with strong reliability and validity. The Pain Disability Index (PDI) will be used to assess the extent to which persistent pain interferes with an individual's ability to engage in seven different areas of everyday activity.
Physical Activity | At baseline, within 1 week prior to surgery, and at 4, 12, and 26 weeks postoperatively.
  Physical activity level will be measured through the Community Health Activities Model Program for Seniors (CHAMPS) questionnaire. In-hospital and in-home physical activity during the acute postoperative period will be measured by the Actiwatch-64, a small wristwatch-like accelerometer device. The Actiwatch will be worn from admission to the in-patient unit until the patient returns to the hospital for catheter removal (approximately 7 days).
Treatment Complications | 26 weeks postoperatively
  The number and type of peri-operative complications will be extracted from medical records.
Length of stay | From time of surgery to discharge (typically 1 week)
  We will collect the postoperative length of stay information for all participants from the patient record.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Derived] Au D, Matthew AG, Lopez P, Hilton WJ, Awasthi R, Bousquet-Dion G, Ladha K, Carli F, Santa Mina D. Prehabilitation and acute postoperative physical activity in patients undergoing radical prostatectomy: a secondary analysis from an RCT. Sports Med Open. 2019 May 22;5(1):18. doi: 10.1186/s40798-019-0191-2. PMID 31119491
- [Derived] Santa Mina D, Matthew AG, Hilton WJ, Au D, Awasthi R, Alibhai SM, Clarke H, Ritvo P, Trachtenberg J, Fleshner NE, Finelli A, Wijeysundera D, Aprikian A, Tanguay S, Carli F. Prehabilitation for men undergoing radical prostatectomy: a multi-centre, pilot randomized controlled trial. BMC Surg. 2014 Nov 13;14:89. doi: 10.1186/1471-2482-14-89. PMID 25394949